CLINICAL TRIAL: NCT04833478
Title: Comparison of Efficacy of Little Lovely Dentist, Dental Song and Tell-show-do Techniques in Alleviating Dental Anxiety in Paediatric Patients -A Single Blind Randomized Controlled Trial
Brief Title: Comparison of Efficacy of Little Lovely Dentist, Dental Song and Tell-show-do Techniques in Alleviating Dental Anxiety in Paediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Hira Abbasi, Principal Investigator, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: Paeds Anxiety
Record Dates: First submitted 2021-03-16; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Anxiety; Paediatric; Dental Anxiety; Behaviour
Keywords: Anxiety; Dental Application; Dental Song; Tell-Show-Do; Behaviour
MeSH Terms: conditions — Anxiety Disorders; Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Application (Experimental): Measuring anxiety level of the patients using Facial Image Scale and Pulse Oximeter
  Interventions: Behavioral: Anxiety
- Dental Song (Experimental): Measuring anxiety level of the patients using Facial Image Scale and Pulse Oximeter
  Interventions: Behavioral: Anxiety
- Tell Show Do (Experimental): Measuring anxiety level of the patients using Facial Image Scale and Pulse Oximeter
  Interventions: Behavioral: Anxiety

INTERVENTIONS:
Behavioral: Anxiety — Techniques used to reduce anxiety in paediatric patients.

SUMMARY:
To evaluate the efficacy of different techniques for the reduction of dental anxiety in pediatric patients. Generally, anxiety amongst paediatric patients is higher as compared to adult patients. So different modalities are used by the dentists in order to reduce the anxiety of such patient to help to make treatment procedures easier and optimal.

DETAILED DESCRIPTION:
Children who suffer from dental anxiety avoid any sort of dental treatment provided to them, which leads to poor oral hygiene, and if unaddressed, problems like missing teeth and decayed teeth further in life develop, and ultimately leading to problems making treatment planning intricate. Children normally follow the footsteps of their parents so it is of importance to consider how to avoid creating dental anxiety among them. If dental anxiety is left untreated, it might persist during adulthood, which eventually will deteriorate the oral health of such patients. Due to the substantial effect of dental anxiety in paediatric patients, many methods have been devised to alleviate or eliminate such anxieties of the patients. This study aimed to employ different strategies and measure heart rate and Facial Image Scale scores to determine their efficacy in reducing paediatric patient's dental anxiety by using these techniques before and after the procedure to compare the effectiveness of each of these techniques.

ELIGIBILITY:
Inclusion Criteria:

* Only the children age ranged from 4 to 11 years with no positive medical history.

Exclusion Criteria:

* Rest were excluded.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Group 1: Little Lovely Dentist App measuring anxiety using pulse oximeter | 5 months
  Measuring Anxiety Levels
Group 1: Little Lovely Dentist App measuring anxiety using facial image scale. | 5 months
  Measuring Anxiety Levels, 1 Minimum value and 5 Maximum value
Group 2: Dental Song measuring anxiety using pulse oximeter | 5 months
  Measuring Anxiety Levels
Group 2: Dental Song measuring anxiety using facial image scale. | 5 months
  Measuring Anxiety Levels, 1 Minimum value and 5 Maximum value
Group 3: Tell-Show-Do measuring anxiety using pulse oximeter | 5 months
  Measuring Anxiety Levels
Group 3: Tell-Show-Do measuring anxiety using facial image scale. | 5 months
  Measuring Anxiety Levels 1 Minimum value and 5 Maximum value

CONTACTS AND LOCATIONS:
Overall Officials: Hira Abbasi, BDS, Post Graduate Trainee, Principal Investigator — Altamash Institute of Dental Medicine
Locations (1):
- Altamash Institute of Dental Medicine, Karachi, Sindh, Pakistan